CLINICAL TRIAL: NCT04157582
Title: Effect of Pilates Training on Cognitive Functions in Patients With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Raghda Nasr Ibrahim Nasr, Assistant Lecturer in Neurological Physical Therapy, October 6 University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 153008
Record Dates: First submitted 2019-10-26; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): will consist of 20 hemiparetic patients and will receive Pilates training in addition to conventional physical therapy program consists of (manual stretching exercises, Strengthening Exercises and Wobble board training ) for 18 sessions every other day for one and half month , 3 sessions /week ,each session for 1.30 hours (40 minutes for pilates then 10 minutes rest then 40 minutes conventional physical therapy).
  Interventions: Other: Pilates training; Other: Conventional physical therapy
- Control group (Experimental): will consist of 20 hemiparetic patients and will receive conventional physical therapy program only same as group I for 18 sessions every other day for one and half month, 3 sessions /week, each session for (40 minutes ).
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Pilates training — 1. Pilates warm-up training (5 minutes) consisted of Breathing, the Chest stretch, the Toy soldier, Upper extremity PNF patterns, and Roll down.
  2. Pilates mat training performed in 5 different positions (30 minutes).
     1. One leg stretch, Hundreds, the Double leg stretch, Scissors, the Shoulder bridge, Oblique preparation, and the Hip twist were performed in the supine position(Fig.7).
     2. Clare, the Side kick, Arm openings, the Lower lift, Leg lifts, and the Side bend were performed in the side-lying position.
     3. Swan dive, the One leg kick, Swimming, the Breast stroke preparations, the Breast stroke performed in the prone position(Fig.8).
     4. Half roll back, Oblique roll up were performed in the sitting position.
     5. Swimming was performed in the kneeling position.
  3. The Pilates cool down training (5 minutes) were the Spine stretch, Saw, Chest stretch, Toy soldier. (Cruz et al .,2011)
  Arms: Study group
Other: Conventional physical therapy — 1. Gentle manual stretching exercises for (elbow flexors, wrist flexors , hamstring and calf muscle).
  2. Strengthening Exercises for ( elbow extensors, wrist extensors and dorsiflexors)
  3. Balance training (Wobble board training) :
     * Patient will stand on squared then circled wobble board while it moves within parallel bars in front of mirror with hand support(with repetition 10times)
     * Patient will stand on squared then circled wobble board while it moves within parallel bars in front of mirror without hand support(with repetition 10times).

SUMMARY:
The purpose of the present study is to investigate the effect of pilates training on cognitive functions in patient with stroke

DETAILED DESCRIPTION:
Stroke remains a primary cause of morbidity throughout the world mainly because of its effect on cognition. Individuals can recover from physical disability resulting from stroke, but might be unable to return to their previous occupations or independent life because of cognitive impairments.

Post-stroke cognitive impairment is not a unitary syndrome but incorporates a variety of deficits in multiple domains such as attention, executive functions , memory, language and visuoperceptual abilities. Cognitive impairment occurs in up to 64% of people who have had a stroke and has been associated with a 3-fold increase in risk for mortality, institutionalization and decreased instrumental activities of daily living function.

Pilates training was developed by Joseph H. Pilates .It belong to a group of so-called Body-Mind Exercises, where the focus is on controlled movement, posture, and breathing .Pilates (pronounced: puh-lah-teez) improves mental and physical well-being , increases flexibility through controlled movements done as mat exercises.

Pilates training improve cognitive functions through increasing blood and oxygen flow to the brain , support neuronal survival in the developping brain ,Generate new neurons ,Provides mood enhancement ,Increases neurotransmitters and Neurotrophins assure the survival of neurons in areas responsible for learning, memory and higher thinking.

ELIGIBILITY:
Inclusion Criteria:

1. Forty patients with stroke (hemiparesis) with muscle power at least grade 3 according to manual muscle testing scale (Appendix VI) from both genders their ages will be ranged from 50-65years old.
2. Patients with ischaemic stroke in the domain of the carotid system.
3. All patients have mild cognitive deficits in domains ( memory, attention, orientation, perception and executive skills) with score <25 according to Montreal Cognitive Assessment (Appendix IV).
4. Duration of illness not less than six months and not more than 18 months.
5. Spastcity grade (1) according to the Modified aschworth scale (MAS) ( Bohannon and Smith, 1987)(Appendix III).
6. All patients in the study should be ambulant independently.
7. Medically and psychologically stable patients.
8. All patients will approve and sign a consent form (Appendix I).
9. All patients are litrate.

Exclusion Criteria:

1. Patients with hemiparesis with motor weakness or incoordination.
2. Patients with cardiovascular problems (uncontrolled hypertension ,unstable angina ,significant coronary heart disease and or congestive heart failure).
3. Patients with dementia with score <3 according to Mini cog test(Appendix V). .
4. Patients with Musculoskeletal problems (deformity or contracture).
5. Medically unstable and uncooperative patients.
6. Patients with Moderate and severe obesity (BMI≥ 35 kg/m2).
7. Patients with depression with score > 8 according to Hamilton depression rating scale (HAM-D) (Appendix VII).

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-10-10 (Estimated); Study Completion 2021-10-20 (Estimated)

PRIMARY OUTCOMES:
Measuring memory function | 45 days
  Vienna test system
Measuring attention | 45 days
  Vienna test system
Measuring orientation | 45 days
  Vienna test system
Measuring perception | 45 days
  Vienna test system
Measuring executive skills | 45 days
  Vienna test system

CONTACTS AND LOCATIONS:
Overall Officials: October 6 University October 6 University, Principal Investigator — October 6 University
Locations (1):
- October 6 university, Giza, Egypt